CLINICAL TRIAL: NCT02014753
Title: Multicenter Comparison of Early and Late Vascular Responses to Everolimus-eluting Cobalt-CHromium Stent and Platelet AggregatioN studIeS for TreatMent of Acute Myocardial Infarction: MECHANISM-AMI
Brief Title: Multicenter Comparison of Early and Late Vascular Responses to Everolimus-eluting Cobalt-CHromium Stent and Platelet AggregatioN studIeS for TreatMent of Acute Myocardial InfarctionTreatment of ST-elevation Acute Myocardial Infarction
Acronym: MECHANISM-AMI
Status: Completed | Type: Observational
Sponsor: Iwate Medical University (Other)
Responsible Party: Principal Investigator, Yoshihiro Morino, Professor, Iwate Medical University
Other Study IDs: MECHANISM-AMI
Record Dates: First submitted 2013-12-12; First posted 2013-12-18 (Estimated); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Coronary Artery Disease
Keywords: AMI; STEMI; ACS
MeSH Terms: conditions — Coronary Artery Disease; ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- CoCr-EES, 2-week OCT follow-up: Undergo primary PCI with cobalt-chromium everolimus-eluting stent (CoCr-EES) for AMI culprit lesion and perform OCT observation at 2-week after PCI.
  Interventions: Device: cobalt-chromium everolimus-eluting stent (CoCr-EES)
- CoCr-EES, 3-month OCT follow-up: Undergo primary PCI with cobalt-chromium everolimus-eluting stent (CoCr-EES) for AMI culprit lesion and perform OCT observation at 3-month after PCI.
  Interventions: Device: cobalt-chromium everolimus-eluting stent (CoCr-EES)

INTERVENTIONS:
Device: cobalt-chromium everolimus-eluting stent (CoCr-EES)
  Other Names: XIENCE PRIME; XIENCE Xpedition

SUMMARY:
To treat patients with acute myocardial infarction, primary percutaneous coronary intervention (PCI) will be performed with the use of an everolimus-eluting cobalt- chromium stent (everolimus-eluting stent: EES, Xience Prime, Xpedition), which is the current standard drug-eluting stent (DES). Vascular responses at the site of stent placement will be evaluated by optical coherence tomography (OCT) at 2 weeks or 3 months and at 12 months after stent placement, along with observation of changes over time in the target vessel. The relationships between OCT findings and the time course of platelet aggregation and between OCT findings and the occurrence of major cardio- cerebrovascular events will also be elucidated.

ELIGIBILITY:
Inclusion Criteria:

- AMI definition is accordance with the third universal definition of ESC /ACCF/ AHA/ WHF Task Force10, detection of a rise and/or fall of cardiac biomarker values [preferably cardiac troponin (cTn) I or T] with at least one value above the 99th percentile upper reference limit (URL) and with at least one of the following: Symptoms of ischemia. New or presumed new significant ST-segment-T wave (ST-T) changes or new left bundlebranch block (LBBB).

Development of pathological Q waves in the ECG. Imaging evidence of new loss of viable myocardium or new regional wall motion abnormality.

Identification of an intracoronary thrombus by angiography or autopsy Of the AMI patients who met the above definition, the criterial for inclusion is limited to STEMI patients. STEMI is defined as new ST elevation at the J point in at least 2 contiguous leads of equal or greater than2 mm (0.2 mV) in men equal or greater than1.5 mm (0.15 mV) in women in leads V2-V3 and/or of equal or greater than 1 mm (0.1 mV) in other contiguous chest leads or the limb leads

* Patients having at least one de novo lesion in a coronary artery in whom PCI with a DES is indicated.
* Patients aged 20 to less than 85 years at the time of informed consent
* Patients who have provided informed consent written by themselves
* Patients who are able to undergo OCT examinations of the site of stent placement at 2 weeks or 3 months and at 12 months.

Exclusion Criteria:

* Shock
* Patients who are judged incapable of undergoing clinical follow-up 12 months after PCI (Consider also the location of patients' residences)
* Lack of specific findings of ACS by angiography (Left to the operator's decision.)
* The culprit lesion is the left main coronary trunk
* Lesion with the reference vascular diameter less than 2.0mm or not less than 4.5mm by visual evaluation.
* Chronic renal failure with serum creatinine level not less than 2.0mg/dl on hospital visit
* Patients on hemodialysis Cancer patients whose vital prognosis is expected to be within 2 years. Surgery that requires discontinuation of the antiplatelet agent is scheduled within 3 months
* Patients who experienced adverse reaction to aspirin or clopidogrel (this shall not apply for patients in whom safety of ticlopidine is confirmed)
* Patients who took warfarin before the onset
* Patients under 20 years old
* Pregnant women
* AMI due to stent thrombosis at prior stented segment.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-04-30 (Actual); Primary Completion 2015-09-25 (Actual); Study Completion 2016-07-26 (Actual)

PRIMARY OUTCOMES:
The percentage of stent strut coverage by OCT | 2 weeks
  To observe temporal course from the early stage, the rate of stent-strut coverage in the 3-months arm will also be evaluated in a complementary manner, separately from the 2-weeks arm.

SECONDARY OUTCOMES:
All-cause Death, Cardiac death, Myocardial Infarction (MI), Stroke, Major bleeding | 1 year
Any Target Lesion Revascularization (TLR) | 1 year
Clinically-driven TLR | 1 year
Any Target Vessel Revascularization (TVR) | 1 year
Coronary-artery bypass surgery (CABG) | 1 year
Any revascularization | 1 year
Angiographic binary restenosis | 1 year
Patient-oriented composite | 1 year
  Composite of All-cause death, any MI including non-target territory, any repeat revascularization and Stroke
OCT Endpoint | 2 weeks and 3 months
  * The percentage of stent strut malapposition
  * The presence of Intra-stent thrombus
  * Intra-stent thrombus area (Maximum site)
  * Intra-stent thrombus length
  * The number of Intra-stent thrombus
Angiographic Quantitative analysis | 12 month
  * In-segment late loss
  * Minimal lumen diameter (MLD), reference vessel diameter (RVD), percent diameter stenosis (%DS)
  * In-stent late loss
  * Binary restenosis (In-stent, In-segment, Peri-stent)
  * Angiographically detected stent fracture（based on Popma's classification ）
  * The number of Intra-stent thrombus
Angiographic Qualitative analysis | 12 month
  * Peri-stent contrast stain (PSS)
  * Site and pattern of restenosis (based on Mehran classification)

OTHER OUTCOMES:
Platelet Aggregation Test | At the time of OCT follow-up (2 weeks or 3 months) and 12 month s
  (1) at the time of PCI, (2) at the time of OCT at 2 weeks or 3 months after PCI, (3) at 12-month follow-up, and (4) at the time of occurrence of a cardio-cerebrovascular event.

CONTACTS AND LOCATIONS:
Locations (1):
- Iwate Medical University Hospital, Morioka, Japan